CLINICAL TRIAL: NCT02406131
Title: Effects of Remote Ischemic Preconditioning on Restenosis Post Lower Limb Revascularization Angioplasty: A Pilot Randomized Control Trial
Brief Title: Effects of Remote Ischemic Preconditioning on Restenosis Post Lower Limb Revascularization Angioplasty
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: logistic issues - no available scans for participants at the moment need to postponed starting dates
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: University College Hospital Galway (Other); University Hospital of Limerick (Other)
Responsible Party: Principal Investigator, KHALID AHMED, Mr, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.A. 1238
Record Dates: First submitted 2015-03-19; First posted 2015-04-02 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Peripheral Vascular Diseases
Keywords: Peripheral Vascular Diseases; Ischemic Preconditioning; Inflammation; Angioplasty; Restenosis; RCT
MeSH Terms: conditions — Peripheral Vascular Diseases; Inflammation

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: (No Intervention): This group will be getting all the routine work up including Duplex scan . we will add request for inflammatory and coagulation markers in their blood samples before and after intervention . The pre-op blood sample will be collected within the 24 hours before intervention and the post intervention in the 24 hrs after (second RIPC window). The repeated duplex scan will be schedule after 6 months.
- RIPC Group (Active Comparator): Remote Ischemic Preconditioning Group (RIPC):This group will have all the tests as for the control group with the additional component will be preconditioning. One hour prior to procedure candidates in this group will have structured intermittent periods of induced remote ischaemic preconditioning using standard blood pressure cuffs. The cuff will be inflated to 200 mmHg applied for 5 minutes alternating with 5 minutes rest to the total of 4 cycles, which needs 40 minutes.
  Interventions: Other: Remote Ischemic Preconditioning

INTERVENTIONS:
Other: Remote Ischemic Preconditioning — standard blood pressure cuffs applied to upper limb . The cuff will be inflated to 200 mmHg applied for 5 minutes alternating with 5 minutes rest to the total of 4 cycles
  Arms: RIPC Group

SUMMARY:
The investigators will established relation between restenosis and inflammatory response to shearing stress caused by angioplasty suggest that any mechanism that affect inflammatory response can consequently affect the restenosis rate. There is accumulated evidence that remote ischemic precondition has modifying suppressive effect on inflammatory response and the investigators hypothesized that RIPC may lead to reduction in post angioplasty restenosis rate.

DETAILED DESCRIPTION:
Rationale:

The father of interventional radiology Charles Dotter (1920-1985) performed the first percutaneous transluminal angioplasty in university of Oregon hospital on Laura Shaw in 16th of January 1964. She presented with typical rest pain and foot gangrene on left leg and her angiogram show distal superficial femoral artery focal stenosis. He saved her leg and she was walking for the next 3 years of her life using his experimental dilating catheter Later in 1977 Zurich witnessed the first coronary angioplasty by German cardiologist Andreas Gruentzig (1939-1985) using same technique .

The angioplasty utilized gradually in the next years after Dotter to provide less invasive option for the growing number of peripheral vascular disease patients estimated to be in the range of 3% to 10%, increasing to 15% to 20% in persons over 70 years. Early diagnosis remains difficult because patients tends to be asymptomatic up to 50% or more of vessel narrowing. the strong association between prevalence of peripheral vascular disease and age increase the demand with world population ageing specially in western Europe and USA. The lower extremity revascularization USA statistics in year 2000 was 40/100,000 and increasing.

Restenosis or the gradual narrowing of the re vascularized vessel remains one of the main problems usually it occurs within 6 months of angioplasty . Restenosis percentages varies between 12% up to 63 % in different studies largely depends on the lesion type and site with below knee interventions being more liable for restenosis.

The restenosis phenomena can be explained by the physiological response to the trauma caused by the balloon when inflated to compress the atheroma. Many factors can influence the process e.g. patient , procedure and vessel condition before intervention.it can be considered as hypertrophic wound healing from the interaction between monocyte-derived macrophages , T cells and arterial wall .the inflammatory response lead to Neointimal Hyperplasia the terminology uses to describe the proliferation and migration of vascular smooth muscle cells . Elevated inflammatory and coagulation factors markers levels after angioplasty has been suggested as predictors for the possibility of restenosis . The inflammatory theory was more supported when using immunosuppressive drugs like Sirolimus shows positive effects on reducing restenosis rate.

Ischemic precondition introduced first as mechanism to reduced subsequent myocardium injury after applying intermittent periods of sub-lethal ischemia . Subsequently the concept examined on other body organs . The mechanisms through which remote ischemic preconditioning (RIPC) work was the subject for many studies suggesting neural, humoral and anti-Inflammatory pathways . Animal studies suggest powerful anti-inflammatory effect for RIPC . other studies shows endothelial protections by decrease formation of reactive oxygen species (ROS) and upregulates endothelial nitric oxide (eNOS) synthase which responsible for most of vasculature Nitric Oxide a very important protective molecule in reperfusion and shearing stress injuries . In human studies Ischaemic, preconditioning show endothelial protective effect and altered Neutrophils function including reduced adhesion, exocytosis, phagocytosis, and modified cytokine secretion. . In one study, RIPC stimulates modified leukocyte inflammatory gene expression in correlations with the first and second windows of the RIPC, which is 1-2 hours and 12-24 respectively.

Sampling Frame the peripheral vascular disease patients with medical profiles, which match trial criteria who are waiting for or admitted from emergency department for lower limb revascularization angioplasty in Galway university hospital, will be identified. Recruitment will be stopped at 10 months of 16 months of the trial period.

Trial Design Patients who need revascularization angioplasty classically had history of symptomatic peripheral vascular disease usually assessed in OPD using ABI and send for duplex ultrasound scan after which some get CT angiogram or Magnetic Resonance Angiography (MRA). Furthermore, intra operative images are the common practice. the investigators will be recruiting from this group in accordance with trial protocol.

The target number will be 40 patients divided into 2 groups. All groups candidates will undergo base line assessment which include history, examination, duplex, ABI and blood sample for inflammatory and coagulation markers.

The candidates will randomly allocated to:

Randomisation Age and DM are associated with many comorbidities. Randomization will be stratified for these two confounders using Minimpy computer software.

All trial candidates will have unique numbers to identify them and conceal their identity. Patients files will be locked in trial office with one-person access and each candidate will get their numbers in sequential way according to their allocation.

Projected recruitment. Galway University hospital provides vascular services for a population of approximately 750000 served by the West-North West Hospitals Group. The patients for the trial will be actively recruited from out patient's clinics, in patients and theatre booking database. Information about the trial will be given to all vascular team including criteria for selection and exclusion. Those who qualified will be counselled by the trial team and consented if the agree to join. The target of 40 patients should be achievable within the recruitment window.

Patient recruitment & consent Eligible candidates will get all the information about the trial in written and verbal explanation for all the steps. Patients who are willing to take part will asked to provide written informed consent. Three copies of the consent form will be signed: one for the patient, one for the patient's clinical notes file and a one copy for the patient's trial folder.

Data collection Demographic and clinical data of eligible candidates who agree to participate will be collected. The candidates will be assign a trial number identifier after informed consent is signed and no personal information will be available on the data entry sheets. The original data-entry preform will be retained together with a copy of the consent form in the trial office with other trial documents in the trial office in CSI building. The code key for the trial numbers will be limited to the Chief Investigator. Encrypted back up copy will be prepared at the end of each data entry and will be kept looked separately. All data will be retained in the care of the principal investigator for a period of five years from the closure of the trial.

Statistical analysis A trial team member blinded to trial allocation will perform the statistical analysis with respect to the primary and secondary outcomes. This is a pilot study the results will be used to identify if there is a need for larger trial.

Trial monitoring Day-to-day management of the trial will be the responsibility of the trial manager, supervised by the principal investigator. A meeting will be held every two weeks between the trial manager and the principal investigator to monitor recruitment, data collection etc.

ELIGIBILITY:
Inclusion criteria

1. Patients planned for lower limb Angioplasty

Exclusion criteria

1. Known upper limb PVD
2. Previous history of upper limb deep vein thrombosis
3. Patients on glibenclamide or nicorandil- May affect RIPC
4. Raynaud's Disease
5. Intra operative decision to use graft - will be documented

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Restenosis | 6 months post procedure
  using Duplex scan 30% stenosis increase in time of flow up. Increase of less than or 50 % stenosis to 70% or more. Loss of 50% of gain in luminal diameter.
Changes in inflammatory and coagulation markers comparing the 2 groups | 24 hours post procedure
  CRP FBC D-Dimer Fibrinogen

SECONDARY OUTCOMES:
Limb Amputation | 6 months post procedure
  recording any limb amputation
Minor amputations | 6 months post procedure
  recording minor amputations - digits
Percentage changes in ABI | 6 months post procedure
  calculate the change in ABI pre and post intervention
Ulcer formation/ healing | 6 months post procedure
  Documents ulcers formation/ healing
Progression of Rutherford classification | 6 months post procedure
  Documents changes pre and post intervention

OTHER OUTCOMES:
Related Data | 6 months post procedure
  Demographic data Smoking DM Lesion type/site Ischemic heart disease Anti- coagulation and Antibiotic usage

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Walsh, Professor, Principal Investigator — NUIGalway - UCHG
Locations (2):
- Ireland (2):
  - University Collage Hospital Galway, Galway, Co Galway
  - Limerick University Hospital, Limerick

REFERENCES:
- [Background] Friedman SG. Charles Dotter and the fiftieth anniversary of endovascular surgery. J Vasc Surg. 2015 Feb;61(2):556-8. doi: 10.1016/j.jvs.2014.09.012. Epub 2014 Oct 11. No abstract available. PMID 25307132
- [Background] Berry D. The unlocking of the coronary arteries: origins of angioplasty. A short historical review of arterial dilatation from Dotter to the creative Gruentzig. Eur Heart J. 2009 Jun;30(12):1421-2. doi: 10.1093/eurheartj/ehp182. No abstract available. PMID 19525552
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). J Vasc Surg. 2007 Jan;45 Suppl S:S5-67. doi: 10.1016/j.jvs.2006.12.037. No abstract available. PMID 17223489
- [Background] Medical Advisory Secretariat. Stenting for peripheral artery disease of the lower extremities: an evidence-based analysis. Ont Health Technol Assess Ser. 2010;10(18):1-88. Epub 2010 Sep 1. PMID 23074395
- [Background] Botev N. Population ageing in Central and Eastern Europe and its demographic and social context. Eur J Ageing. 2012 Feb 9;9(1):69-79. doi: 10.1007/s10433-012-0217-9. eCollection 2012 Mar. PMID 28804408
- [Background] Anderson PL, Gelijns A, Moskowitz A, Arons R, Gupta L, Weinberg A, Faries PL, Nowygrod R, Kent KC. Understanding trends in inpatient surgical volume: vascular interventions, 1980-2000. J Vasc Surg. 2004 Jun;39(6):1200-8. doi: 10.1016/j.jvs.2004.02.039. PMID 15192558
- [Background] Nowygrod R, Egorova N, Greco G, Anderson P, Gelijns A, Moskowitz A, McKinsey J, Morrissey N, Kent KC. Trends, complications, and mortality in peripheral vascular surgery. J Vasc Surg. 2006 Feb;43(2):205-16. doi: 10.1016/j.jvs.2005.11.002. PMID 16476588
- [Background] Serruys PW, Luijten HE, Beatt KJ, Geuskens R, de Feyter PJ, van den Brand M, Reiber JH, ten Katen HJ, van Es GA, Hugenholtz PG. Incidence of restenosis after successful coronary angioplasty: a time-related phenomenon. A quantitative angiographic study in 342 consecutive patients at 1, 2, 3, and 4 months. Circulation. 1988 Feb;77(2):361-71. doi: 10.1161/01.cir.77.2.361. PMID 2962786
- [Background] Schillinger M, Exner M, Mlekusch W, Haumer M, Rumpold H, Ahmadi R, Sabeti S, Wagner O, Minar E. Endovascular revascularization below the knee: 6-month results and predictive value of C-reactive protein level. Radiology. 2003 May;227(2):419-25. doi: 10.1148/radiol.2272020137. Epub 2003 Mar 20. PMID 12649419
- [Background] Cejna M, Thurnher S, Illiasch H, Horvath W, Waldenberger P, Hornik K, Lammer J. PTA versus Palmaz stent placement in femoropopliteal artery obstructions: a multicenter prospective randomized study. J Vasc Interv Radiol. 2001 Jan;12(1):23-31. doi: 10.1016/s1051-0443(07)61397-9. PMID 11200349
- [Background] Tsigkas GG, Karantalis V, Hahalis G, Alexopoulos D. Stent restenosis, pathophysiology and treatment options: a 2010 update. Hellenic J Cardiol. 2011 Mar-Apr;52(2):149-57. No abstract available. PMID 21478125
- [Background] Schillinger M, Minar E. Restenosis after percutaneous angioplasty: the role of vascular inflammation. Vasc Health Risk Manag. 2005;1(1):73-8. doi: 10.2147/vhrm.1.1.73.58932. PMID 17319099
- [Background] Kleinedler JJ, Foley JD, Orchard EA, Dugas TR. Novel nanocomposite stent coating releasing resveratrol and quercetin reduces neointimal hyperplasia and promotes re-endothelialization. J Control Release. 2012 Apr 10;159(1):27-33. doi: 10.1016/j.jconrel.2012.01.008. Epub 2012 Jan 17. PMID 22269665
- [Background] Wahlgren CM, Sten-Linder M, Egberg N, Kalin B, Blohme L, Swedenborg J. The role of coagulation and inflammation after angioplasty in patients with peripheral arterial disease. Cardiovasc Intervent Radiol. 2006 Jul-Aug;29(4):530-5. doi: 10.1007/s00270-005-0159-0. PMID 16729229
- [Background] Tschopl M, Tsakiris DA, Marbet GA, Labs KH, Jager K. Role of hemostatic risk factors for restenosis in peripheral arterial occlusive disease after transluminal angioplasty. Arterioscler Thromb Vasc Biol. 1997 Nov;17(11):3208-14. doi: 10.1161/01.atv.17.11.3208. PMID 9409313
- [Background] Hausleiter J, Kastrati A, Mehilli J, Vogeser M, Zohlnhofer D, Schuhlen H, Goos C, Pache J, Dotzer F, Pogatsa-Murray G, Dirschinger J, Heemann U, Schomig A; OSIRIS Investigators. Randomized, double-blind, placebo-controlled trial of oral sirolimus for restenosis prevention in patients with in-stent restenosis: the Oral Sirolimus to Inhibit Recurrent In-stent Stenosis (OSIRIS) trial. Circulation. 2004 Aug 17;110(7):790-5. doi: 10.1161/01.CIR.0000138935.17503.35. Epub 2004 Aug 9. PMID 15302787
- [Background] Murry CE, Jennings RB, Reimer KA. Preconditioning with ischemia: a delay of lethal cell injury in ischemic myocardium. Circulation. 1986 Nov;74(5):1124-36. doi: 10.1161/01.cir.74.5.1124. PMID 3769170
- [Background] Przyklenk K, Bauer B, Ovize M, Kloner RA, Whittaker P. Regional ischemic 'preconditioning' protects remote virgin myocardium from subsequent sustained coronary occlusion. Circulation. 1993 Mar;87(3):893-9. doi: 10.1161/01.cir.87.3.893. PMID 7680290
- [Background] Jensen HA, Loukogeorgakis S, Yannopoulos F, Rimpilainen E, Petzold A, Tuominen H, Lepola P, Macallister RJ, Deanfield JE, Makela T, Alestalo K, Kiviluoma K, Anttila V, Tsang V, Juvonen T. Remote ischemic preconditioning protects the brain against injury after hypothermic circulatory arrest. Circulation. 2011 Feb 22;123(7):714-21. doi: 10.1161/CIRCULATIONAHA.110.986497. Epub 2011 Feb 7. PMID 21300953
- [Background] Wang Y, Shen J, Xiong X, Xu Y, Zhang H, Huang C, Tian Y, Jiao C, Wang X, Li X. Remote ischemic preconditioning protects against liver ischemia-reperfusion injury via heme oxygenase-1-induced autophagy. PLoS One. 2014 Jun 10;9(6):e98834. doi: 10.1371/journal.pone.0098834. eCollection 2014. PMID 24914543
- [Background] Hausenloy DJ, Yellon DM. Remote ischaemic preconditioning: underlying mechanisms and clinical application. Cardiovasc Res. 2008 Aug 1;79(3):377-86. doi: 10.1093/cvr/cvn114. Epub 2008 May 2. PMID 18456674
- [Background] Souza Filho MV, Loiola RT, Rocha EL, Simao AF, Gomes AS, Souza MH, Ribeiro RA. Hind limb ischemic preconditioning induces an anti-inflammatory response by remote organs in rats. Braz J Med Biol Res. 2009 Oct;42(10):921-9. doi: 10.1590/s0100-879x2009005000025. Epub 2009 Sep 11. PMID 19738981
- [Background] Zhang JQ, Wang Q, Xue FS, Li RP, Cheng Y, Cui XL, Liao X, Meng FM. Ischemic preconditioning produces more powerful anti-inflammatory and cardioprotective effects than limb remote ischemic postconditioning in rats with myocardial ischemia-reperfusion injury. Chin Med J (Engl). 2013 Oct;126(20):3949-55. PMID 24157164
- [Background] Kim YH, Yoon DW, Kim JH, Lee JH, Lim CH. Effect of remote ischemic post-conditioning on systemic inflammatory response and survival rate in lipopolysaccharide-induced systemic inflammation model. J Inflamm (Lond). 2014 May 21;11:16. doi: 10.1186/1476-9255-11-16. eCollection 2014. PMID 24904237
- [Background] He X, Zhao M, Bi XY, Yu XJ, Zang WJ. Delayed preconditioning prevents ischemia/reperfusion-induced endothelial injury in rats: role of ROS and eNOS. Lab Invest. 2013 Feb;93(2):168-80. doi: 10.1038/labinvest.2012.160. Epub 2012 Nov 12. PMID 23147223
- [Background] Roviezzo F, Cuzzocrea S, Di Lorenzo A, Brancaleone V, Mazzon E, Di Paola R, Bucci M, Cirino G. Protective role of PI3-kinase-Akt-eNOS signalling pathway in intestinal injury associated with splanchnic artery occlusion shock. Br J Pharmacol. 2007 Jun;151(3):377-83. doi: 10.1038/sj.bjp.0707233. Epub 2007 Apr 23. PMID 17450173
- [Background] Forstermann U, Munzel T. Endothelial nitric oxide synthase in vascular disease: from marvel to menace. Circulation. 2006 Apr 4;113(13):1708-14. doi: 10.1161/CIRCULATIONAHA.105.602532. PMID 16585403
- [Background] Shimizu M, Saxena P, Konstantinov IE, Cherepanov V, Cheung MM, Wearden P, Zhangdong H, Schmidt M, Downey GP, Redington AN. Remote ischemic preconditioning decreases adhesion and selectively modifies functional responses of human neutrophils. J Surg Res. 2010 Jan;158(1):155-61. doi: 10.1016/j.jss.2008.08.010. PMID 19540519
- [Background] Kharbanda RK, Peters M, Walton B, Kattenhorn M, Mullen M, Klein N, Vallance P, Deanfield J, MacAllister R. Ischemic preconditioning prevents endothelial injury and systemic neutrophil activation during ischemia-reperfusion in humans in vivo. Circulation. 2001 Mar 27;103(12):1624-30. doi: 10.1161/01.cir.103.12.1624. PMID 11273988
- [Background] Konstantinov IE, Arab S, Kharbanda RK, Li J, Cheung MM, Cherepanov V, Downey GP, Liu PP, Cukerman E, Coles JG, Redington AN. The remote ischemic preconditioning stimulus modifies inflammatory gene expression in humans. Physiol Genomics. 2004 Sep 16;19(1):143-50. doi: 10.1152/physiolgenomics.00046.2004. Epub 2004 Aug 10. PMID 15304621
- [Background] Hausenloy DJ, Yellon DM. The second window of preconditioning (SWOP) where are we now? Cardiovasc Drugs Ther. 2010 Jun;24(3):235-54. doi: 10.1007/s10557-010-6237-9. PMID 20496105
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250